CLINICAL TRIAL: NCT05800977
Title: A Phase 1b/2 Study of a Anti-CD19/CD20 Bispecific CAR-T Therapy (C-CAR039/Prizloncabtagene Autoleucel) in Patients With Relapsed/Refractory Large B-Cell Lymphoma
Brief Title: A Study of C-CAR039 (Prizloncabtagene Autoleucel) in Patients With Relapsed/Refractory Large B-Cell Lymphoma
Acronym: ELEVATION
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-032
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Large B-Cell Lymphoma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prizloncabtagene Autoleucel (Experimental): Prizlon-cel will be intravenously administered as a single infusion after lymphodepletion.
  Interventions: Biological: Prizloncabtagene autoleucel

INTERVENTIONS:
Biological: Prizloncabtagene autoleucel — Prizlon-cel is a novel 2nd generation 4-1BB bispecific chimeric antigen receptor T-cell (CAR-T) targeting both CD19 and CD20 antigens
  Other Names: C-CAR039

SUMMARY:
This is a multicenter, single arm, open-label study. The purpose of the study is to evaluate safety of Prizloncabtagene Autoleucel (Prizlon-cel) and establish the recommended Phase 2 dose (RP2D) (Phase 1b) and to evaluate the efficacy of Prizlon-cel (Phase 2) in patients with relapsed or refractory large b-cell lymphoma (LBCL).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and efficacy of Prizlon-cel. It includes two phases, Phase 1b and Phase 2. In Phase 1b study, RP2D will be determined. The selected dose will be further evaluated in the Phase 2 study. The study includes the following sequential procedures: Screening, Apheresis and CAR-T manufacturing, Baseline, Lymphodepletion, CAR-T infusion, DLT period (Phase 1b) and Follow-up Visit. Subjects will be followed for at least 2 years after Prizlon-cel infusion, with up to 15 years long-term follow-up on a separate study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically confirmed CD19 or CD20 positive B-cell non-Hodgkin lymphoma, including the following neoplasms as defined by the 2016 WHO classification of lymphoid neoplasms:

  1. Diffuse large B-cell lymphoma, not otherwise specified (DLBCL, NOS)
  2. Primary mediastinal large B-cell lymphoma (PMBCL)
  3. Transformed follicular lymphoma (tFL)
  4. High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements (HGBL-DH/TH)
  5. High-grade B-cell lymphoma, NOS (HGBL, NOS)
  6. Follicular lymphoma grade 3B (FL3B)
* Relapsed or refractory disease after ≥ 2 lines of standard therapy or relapsed after autologous stem cell transplantation (ASCT)
* At least one measurable lesion per the Lugano 2014 Classification
* Adequate organ and marrow function

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplantation (HSCT) at anytime, or ASCT within 12 weeks prior to apheresis
* Suspected or confirmed central nervous system involvement
* Stroke or convulsion history within 6 months of signing informed consent form (ICF)
* Autoimmune disease, immunodeficiency or diseases requiring immunosuppressants treatment
* Uncontrolled active infection
* Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA in peripheral blood; positive hepatitis C virus (HCV) antibody with positive HCV RNA in peripheral blood; positive human immunodeficiency virus (HIV) antibody; positive syphilis test
* Severe heart, liver, renal or metabolism disease
* Inadequate wash-out time for previous anti-tumor treatments prior to apheresis
* Prior CAR-T therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Incidence and Severity of Treatment-emergent Adverse Events (TEAEs) | Up to 90 days after C-CAR039 infusion
  Incidence and severity of TEAEs , including dose limiting toxicities (DLTs)
Phase 1b: Recommended Phase 2 Dose (R2PD) | Up to 3 months after C-CAR039 infusion
  Based on DLTs rates and overall safety profile
Phase 2: Overall Response Rate (ORR) at 3 months | Up to 3 months after C-CAR039 infusion
  Best response rate at 3 months after C-CAR039 infusion, including partial response (PR) and complete response (CR)

SECONDARY OUTCOMES:
Phase 1b: Incidence and Severity of Adverse Events (AEs) | Up to 2 years after C-CAR039 infusion
  Incidence and severity of AEs
Phase 1b: ORR at 3 months | Up to 3 months after C-CAR039 infusion
  Best response rate at 3 months after C-CAR039 infusion, including PR and CR
Phase 2: Incidence and Severity of Adverse Events (AEs) | Up to 2 years after C-CAR039 infusion
  Incidence and severity of any AEs
ORR | Up to 2 years after C-CAR039 infusion
  Best response, including PR and CR
ORR at 6 months | Up to 6 months after C-CAR039 infusion
  Best response rate at 6 months after C-CAR039 infusion, including PR and CR
Duration of response (DOR) | Up to 2 years after C-CAR039 infusion
  The time from the first documented PR or CR to disease progression or death, whichever occurs first
Time to response (TTR) | Up to 2 years after C-CAR039 infusion
  The time from the date of C-CAR039 infusion to the first documented PR or CR
Progression-free survival (PFS) | Up to 2 years after C-CAR039 infusion
  The time from the date of C-CAR039 infusion to the date of first documented disease progression or death
Overall survival (OS) | Up to 2 years after C-CAR039 infusion
  The time from the date of C-CAR039 infusion to the date of death
Maximal plasma concentration (Cmax) | Up to 2 years after C-CAR039 infusion
  Maximal plasma concentration of C-CAR039 in peripheral blood
Time to reach the maximal plasma concentration (Tmax) | Up to 2 years after C-CAR039 infusion
  Time to reach the maximal plasma concentration of C-CAR039 in peripheral blood
Area under the curve within 28 days (AUC0-28d) | Up to 28 days after C-CAR039 infusion
  Area under the curve of C-CAR039 in peripheral blood within 28 days post infusion
Time of last measurable observed concentration (Tlast) | Up to 2 years after C-CAR039 infusion
  Time of last measurable observed concentration of C-CAR039 in peripheral blood
The B cell percentage changes and CD19/CD20 expression changes in blood | Up to 2 years after C-CAR039 infusion
  The B cell percentage changes and CD19/CD20 expression changes in blood by flow cytometry assay before and after C-CAR039 infusion
Anti-drug (C-CAR039) antibody | Up to 2 years after C-CAR039 infusion
  Presence of serum anti-drug (C-CAR039) antibody

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, M.D., PhD, Principal Investigator — Ruijin Hospital; Lugui Qiu, Principal Investigator — Chinese Academy of Medical Sciences Hematology Hospital
Locations (15):
- China (15):
  - Beijing Cancer Hospital, Beijing
  - Beijing GoBroad Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Jiangxi Cancer Hospital, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Chinese Academy of Medical Sciences Hematology Hospital, Tianjin
  - Tianjin Medical University Cancer Institute& Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No